CLINICAL TRIAL: NCT03848312
Title: Cognitive Training to Reduce Incidence of Cognitive Impairment in Older Adults
Brief Title: Preventing Alzheimer's With Cognitive Training
Acronym: PACT
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University of South Florida (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Jennifer L. O'Brien, Associate Professor, University of South Florida
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: WIRB® Protocol #20182630; 1R56AG058234-01A1 (NIH); 1R01AG070349-01 (NIH)
Record Dates: First submitted 2019-02-14; First posted 2019-02-20 (Actual); Last update posted 2024-09-26 (Actual); Status verified 2024-09

CONDITIONS: Age-related Cognitive Decline; Alzheimer's Disease and Related Dementias
MeSH Terms: conditions — Alzheimer Disease | interventions — Cognitive Training

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Computerized Cognitive Training (Experimental): Participants will complete computerized cognitive training.
  Interventions: Behavioral: Cognitive Training
- Computerized Cognitive Stimulation (Active Comparator): Participants will complete cognitively-stimulating computer activities.
  Interventions: Behavioral: Computerized Cognitive Stimulation

INTERVENTIONS:
Behavioral: Cognitive Training — Participants will be completing a total of 45 computerized sessions.
  Arms: Computerized Cognitive Training
Behavioral: Computerized Cognitive Stimulation — Participants will be completing a total of 45 computerized cognitive stimulation sessions.
  Arms: Computerized Cognitive Stimulation

SUMMARY:
Dementia is the most expensive medical condition in the US and increases in prevalence with age. More than 5 million Americans have Alzheimer's disease, the most common form of dementia. Mild cognitive impairment is a transitional stage between normal cognitive aging and Alzheimer's disease or another type of dementia, and is indicative of higher risk for dementia. In addition to the obvious health and quality-of-life ramifications of dementia, there are high direct (e.g., subsidizing residential care needs) and indirect (e.g., lost productivity of family caregivers) economic costs. Implementing interventions to prevent MCI and dementia among older adults is of critical importance to health and maintained quality-of-life for millions of Americans. Recent data analyses from the Advanced Cognitive Training in Vital Elderly study (ACTIVE) indicate that a specific cognitive intervention, speed of processing training (SPT), significantly delays the incidence of cognitive impairment across 10 years. The primary contribution of the proposed research will be the determination of whether this cognitive training technique successfully delays the onset of clinically defined MCI or dementia across three years.

DETAILED DESCRIPTION:
Preventing Alzheimer's Disease with Cognitive Training: The PACT Trial

The primary objective in the R56 phase was to establish the feasibility of the proposed field trial including meeting participant enrollment goals. The feasibility of the field trial was established by accruing 1000 enrolled participants. The secondary objective in the R56 phase was to ascertain participants' willingness to enroll in a longitudinal clinical trial and to subsequently complete a multispecialty clinical diagnostic evaluation, psychometric testing, MRI, PET scan, and genetic testing. Participants' willingness to allow access to medicare records was also determined.

The trial is being expanded in the R01 phase with the goal of enrolling 7600 participants.

The primary goal is to ascertain the effectiveness of cognitive speed of processing training (SPT) to reduce the incidence of Mild Cognitive Impairment (MCI) or dementia.

Design and Outcomes: A randomized clinical trial among 7600 adults 65 years of age and older will be completed in order to test the effectiveness of computerized cognitive speed of processing training (SPT) to reduce incidence of MCI or dementia.

Participants will be screened with an inclusion/exclusion questionnaire and those potentially eligible will complete brief memory screening, depression screening, and other questionnaires. Those eligible will be randomized to one of two conditions of brain games and will complete at least two in-person, supervised training sessions. Additional exercises will be completed at-home over the next 3 to 5 months followed by booster sessions 1- and 2-years later.

Participants are asked to initially complete 25 sessions of training and will be asked complete an additional 10 sessions of booster training 1- and 2- years later. Participants are instructed to complete 2-3 sessions of training per week until 25 sessions are completed. At 1- year and again at 2-years, participants will be instructed to complete an additional 10 sessions of training.

Sample Size and Population: Adults 65 years of age and older (N=7600) will be randomly assigned to SPT (n=3800) or the active comparator condition (n=3800).

ELIGIBILITY:
Inclusion Criteria:

* Be age 65 or older at time of consent
* Have ability to speak and understand English or Spanish
* Report adequate sensorimotor capacity to perform the computer exercises
* Report adequate visual capacity to read from a computer screen at a typical viewing distance
* Show adequate auditory capacity to understand conversational speech
* Show adequate motor capacity to touch a computer screen or control a computer mouse.
* Have no evidence of Mild Cognitive Impairment (MCI) or dementia, as assessed by the Montreal Cognitive Assessment score >=26.
* Have adequate mental health (no self-reported diagnoses of mental illness that would interfere with ability to comply with study procedures or benefit from intervention)
* Wiling to complete all study activities
* Ability to understand study procedures and comply with them for the length of the study

Exclusion Criteria:

* Currently enrolled in another randomized clinical trial, treatment trial, or another research study that assesses cognition
* Previous participation in a cognitive training study
* Self-reported vision, hearing, or motor difficulties that would interfere with the ability to complete the study interventions
* Self-reported diagnosis of mild cognitive impairment, dementia, stroke, traumatic brain injury, brain tumor, or a neurological disorder that affects cognition or would interfere with the ability to benefit from the study intervention (e.g., Parkinson disease, multiple sclerosis), or any other unstable medical conditions that is predisposing to imminent cognitive or functional decline (e.g., congestive heart failure, chronic obstructive pulmonary disorder dependent on oxygen, or undergoing chemotherapy or radiation).
* Self-reported use of medications typically prescribed for dementia such as: Namenda, Memantine, Namzaric, Donepezil, Aricept, Rivastigmine, Exelon, Razadyne, Galantamine, Reminyl, aducanumab, Aduhlem.
* Completion of 10 or more hours of a computerized cognitive training program in the last 5 years such as: Lumosity, Posit Science Brain Fitness, InSight, or Brain HQ, Lace, CogMed, CogniFit, Happy Neuron, Elevate, or Dakim
* Severe depressive symptoms (Geriatric Depression Scale score >=5)

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 7600 (Estimated)
Dates: Start 2019-02-19 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of mild cognitive impairment or dementia | Three years
  clinical diagnosis of mild cognitive impairment or dementia

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - University of Florida, Gainesville, Florida
  - University of Florida, Jacksonville, Florida
  - University of North Florida, Jacksonville, Florida
  - The Roskamp Institute, Sarasota, Florida
  - University of South Florida, Tampa, Florida
  - Duke Health, Durham, North Carolina
  - Clemson University Institute for Engaged Aging, Seneca, South Carolina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nicholson JS, Hudak EM, Phillips CB, Chanti-Ketterl M, O'Brien JL, Ross LA, Lister JJ, Burke JR, Potter G, Plassman BL, Woods AJ, Krischer J, Edwards JD. The Preventing Alzheimer's with Cognitive Training (PACT) randomized clinical trial. Contemp Clin Trials. 2022 Dec;123:106978. doi: 10.1016/j.cct.2022.106978. Epub 2022 Oct 28. PMID 36341846

DOCUMENTS (1):
  • Statistical Analysis Plan (2019-11-04): https://cdn.clinicaltrials.gov/large-docs/12/NCT03848312/SAP_000.pdf